CLINICAL TRIAL: NCT04669899
Title: Phase 1/2 First-in-Human (FIH) Study of Leukocyte Immunoglobulin-Like Receptor B2 (LILRB2) Inhibitor Monoclonal Antibody (mAb) JTX-8064, as Monotherapy and in Combination With a Programmed Cell Death Receptor-1 (PD-1) Inhibitor, in Adult Subjects With Advanced Refractory Solid Tumor Malignancies
Brief Title: Study of JTX-8064, as Monotherapy and in Combination With a PD-1 Inhibitor, in Adult Subjects With Advanced Refractory Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jounce Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JTX-8064-101
Record Dates: First submitted 2020-12-04; First posted 2020-12-17 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Cancer
Keywords: JTX-8064; LILRB2; ILT4; PD-1; JTX-4014; Immunotherapy; Immuno-oncology; Solid tumor Malignancies; Dose escalation; INNATE; Monotherapy; Combination Therapy; Antineoplastic Agents; Immunological
MeSH Terms: conditions — Neoplasms | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Stage 1, Dose Escalation: JTX-8064 monotherapy dose escalation (Experimental): Dose Escalation, Stage 1: JTX-8064 Monotherapy. Cohorts will enroll subjects with histologically or cytologically confirmed advanced/metastatic extracranial solid tumor malignancies.
  Interventions: Drug: JTX-8064
- Stage 2, Dose Escalation: JTX-8064 in combination with pimivalimab (Experimental): Dose Escalation, Stage 2: JTX-8064 in combination with pimivalimab. Cohorts will enroll subjects with histologically or cytologically confirmed advanced/metastatic extracranial solid tumor malignancies.
  Interventions: Drug: JTX-8064; Drug: pimivalimab
- Stage 3 Expansion: JTX-8064 monotherapy (Ovarian) (Experimental): Cohort will enroll subjects with advanced/metastatic PD-1/PD-L1 (PD-(L)1)-naïve, platinum-resistant ovarian cancer.
  Interventions: Drug: JTX-8064
- Stage 4, Expansion: JTX-8064 in combination with pimivalimab (ccRCC) (Experimental): JTX-8064 in combination with pimivalimab. Cohort will enroll subjects with advanced/metastatic PD-(L)1i-experienced clear cell renal cell carcinoma (ccRCC).
  Interventions: Drug: JTX-8064; Drug: pimivalimab
- Stage 4, Expansion: JTX-8064 in combination with pimivalimab (TNBC) (Experimental): JTX-8064 in combination with pimivalimab. Cohort will enroll subjects with advanced/metastatic PD-(L)1i-experienced triple negative breast cancer (TNBC).
  Interventions: Drug: JTX-8064; Drug: pimivalimab
- Stage 4, Expansion: JTX-8064 in combination with pimivalimab (HNSCC) (Experimental): JTX-8064 in combination with pimivalimab. Cohort will enroll subjects with advanced/metastatic PD-(L)1-naïve, PD-L1+ head and neck squamous cell carcinoma (HNSCC).
  Interventions: Drug: JTX-8064; Drug: pimivalimab
- Stage 4, Expansion: JTX-8064 in combination with pimivalimab (Ovarian) (Experimental): JTX-8064 in combination with pimivalimab. Cohort will enroll subjects with advanced/metastatic PD-(L)1-naïve, platinum-resistant ovarian cancer.
  Interventions: Drug: JTX-8064; Drug: pimivalimab
- Stage 4, Expansion: JTX-8064 in combination with pimivalimab (NSCLC) (Experimental): JTX-8064 in combination with pimivalimab. Cohort will enroll subjects with advanced/metastatic PD-(L)1-experienced non-small cell lung cancer (NSCLC).
  Interventions: Drug: JTX-8064; Drug: pimivalimab
- Stage 4, Expansion: JTX-8064 in combination with pimivalimab (cSCC) (Experimental): JTX-8064 in combination with pimivalimab. Cohort will enroll subjects with advanced/metastatic PD-(L)1-experienced cutaneous squamous cell carcinoma (cSCC).
  Interventions: Drug: JTX-8064; Drug: pimivalimab
- Stage 4, Expansion: JTX-8064 in combination with pimivalimab (UPS & LPS) (Experimental): JTX-8064 in combination with pimivalimab. Cohort will enroll subjects with advanced/metastatic PD-(L)1-naïve undifferentiated pleomorphic sarcoma (UPS) and liposarcoma (LPS).
  Interventions: Drug: JTX-8064; Drug: pimivalimab
- Stage 4, Expansion: JTX-8064 in combination with pimivalimab (PD-(L)1i-experienced HNSCC) (Experimental): JTX-8064 in combination with pimivalimab. Cohort will enroll subjects with PD-(L)1i-experienced HNSCC.
  Interventions: Drug: JTX-8064; Drug: pimivalimab
- Stage 4, Expansion: JTX-8064 in combination with pimivalimab (BTC) (Experimental): JTX-8064 in combination with pimivalimab. Cohort will enroll subjects with biliary tract cancer (BTC), including intra-and extra-hepatic biliary duct cancer and cancer of the gallbladder. All subjects must have progressed on or after gemcitabine/cisplatin (Gem/Cis) in the metastatic setting, must have PD-(L)1i resistance.
  Interventions: Drug: JTX-8064; Drug: pimivalimab

INTERVENTIONS:
Drug: JTX-8064 — Specified dose on specified days
  Other Names: Anti-LILRB2; Anti-ILT4
Drug: pimivalimab — Specified dose on specified days
  Other Names: JTX-4014; Anti-PD-1
  Arms: Stage 2, Dose Escalation: JTX-8064 in combination with pimivalimab; Stage 4, Expansion: JTX-8064 in combination with pimivalimab (BTC); Stage 4, Expansion: JTX-8064 in combination with pimivalimab (HNSCC); Stage 4, Expansion: JTX-8064 in combination with pimivalimab (NSCLC); Stage 4, Expansion: JTX-8064 in combination with pimivalimab (Ovarian); Stage 4, Expansion: JTX-8064 in combination with pimivalimab (PD-(L)1i-experienced HNSCC); Stage 4, Expansion: JTX-8064 in combination with pimivalimab (TNBC); Stage 4, Expansion: JTX-8064 in combination with pimivalimab (UPS & LPS); Stage 4, Expansion: JTX-8064 in combination with pimivalimab (cSCC); Stage 4, Expansion: JTX-8064 in combination with pimivalimab (ccRCC)

SUMMARY:
JTX-8064-101 is a Phase 1/2, open label, dose escalation and dose expansion clinical study to determine the safety, tolerability, and recommended Phase 2 dose (RP2D) of JTX-8064 alone and in combination with a PD-1 inhibitor (PD-1i).

DETAILED DESCRIPTION:
JTX-8064 is a humanized mAb designed to block the interaction of LILRB2 with its known ligands, endogenous major histocompatibility complex class I (MHC I) molecules. This is a Phase 1/2, first in human, open label, multicenter, dose escalation and dose expansion clinical trial to determine the safety, tolerability, maximum tolerated dose (MTD) and RP2D of JTX-8064 when administered as a single agent and in combination with a PD-1i in adult subjects with advanced refractory solid tumor malignancies. Additionally, the study will seek to evaluate the pharmacokinetics and immunogenicity of JTX-8064, and preliminary efficacy of JTX-8064 as a monotherapy and in combination with a PD-1i.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to participate and comply with all study requirements and provide signed and dated informed consent prior to initiation of any study procedures;
2. Histologically or cytologically confirmed advanced/metastatic extracranial solid tumor malignancy:

   1. Stages 1 and 2: Subjects must have received, have been intolerant to, have been ineligible for, or have declined all treatment known to confer clinical benefit with the exception of subjects enrolled in combination cohorts with a PD-1i, where a PD-1i is approved by the local regulatory agencies;
   2. Stage 3: This stage may enroll subjects with 3L/4L PD-(L)1-naïve, platinum-resistant ovarian cancer;
   3. Stage 4: This stage may enroll subjects with the following cancers:

      * 2L/3L ccRCC. Subjects must have progressed on or after treatment with an anti-PD-(L)1 agent in their most recent prior line of therapy;
      * 2L-4L TNBC. Subjects must have progressed on or after treatment with a prior anti-PD-(L)1 therapy;
      * 1L, PD-(L)1-naïve, PD-L1+; combined positive score (CPS) ≥1% HNSCC;
      * 2L/3L platinum-experienced HNSCC. Subjects must have progressed on or after treatment with an anti-PD-(L)1-agent in their most recent prior line of therapy;
      * 3L/4L, PD-(L)1-naïve, platinum-resistant ovarian cancer;
      * 2L/3L NSCLC. Subjects must have progressed on or after treatment with platinum-based chemotherapy and an anti-PD-(L)1-containing therapy. The anti-PD-(L)1 agent must have been a part of the most recent prior line of therapy. Subjects with EGFR mutations and ALK rearrangements will be excluded. Subjects with other targetable genomic aberrations for which FDA approved therapies exist must have received appropriate FDA-approved targeted therapy;
      * 2L/3L cSCC. Subjects must have progressed on or after treatment with an anti-PD-(L)1 agent in their most recent prior line of therapy;
      * 2L-4L PD-(L)1-naïve undifferentiated pleomorphic sarcoma (UPS) and liposarcoma (LPS);
      * 2L/3L biliary tract cancer (BTC), including intra- and extra-hepatic biliary duct cancer and cancer of the gallbladder. Subjects must have progressed on or after gemcitabine/cisplatin (Gem/Cis) in the metastatic setting and must have PD-(L)1 inhibitor resistance. Subjects with FGFR and IDH1 mutations must have progressed on or after targeted therapies for these mutations;
3. Measurable disease, according to the RECIST version 1.1, that has objectively progressed since (or on) previous treatment as assessed by the Investigator;
4. ≥18 years of age;
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
6. Predicted life expectancy of ≥3 months;
7. Have specified laboratory values (obtained ≤28 days prior to planned Cycle 1, Day 1 [C1D1]) in accordance with the study protocol;
8. For women of childbearing potential (WOCBP): negative serum pregnancy test during the Screening period and a negative urine pregnancy test up to 24 hours in advance of C1D1;
9. WOCBP and males whose partners are WOCBP must agree to use a highly effective method of birth control throughout their participation and for 5 months following the last study drug administration.

Exclusion Criteria:

1. Concurrent anticancer treatment, either FDA approved or investigational, for the cancer being evaluated in this study or for prior malignancies. A past history of other malignancies is allowed as long as the subject is not receiving treatment other than hormonal therapy and, in the judgment of the Investigator, is unlikely to have a recurrence. Of note, concurrent malignancies that do not require treatment and are clinically stable are allowed;
2. Prior infusion of JTX-8064, LILRB2, or ILT4-directed therapy;
3. The therapies listed below within the specified timeframe or ongoing toxicity attributed to prior therapy that was >Grade 1 according to the NCI CTCAE, version 5.0. Exceptions: >Grade 1 toxicities that, in the opinion of the Investigator, should not exclude the subject (e.g., alopecia, Grade 2 neuropathy, hypo- or hyperthyroidism, or other endocrinopathies that are well controlled with hormone replacement) and are approved by the Medical Monitor:

   1. Major surgery (excluding minor procedures, for example, placement of vascular access, gastrointestinal/biliary stent, biopsy) <4 weeks prior to planned C1D1;
   2. Immunotherapy or biologic therapy <28 days prior to planned C1D1 or 5 half-lives, whichever is shorter;
   3. Chemotherapy <21 days prior to planned C1D1, or <42 days for mitomycin or nitrosoureas or 5 half-lives, whichever is shorter;
   4. Targeted small molecule therapy <14 days or 5 half-lives, whichever is shorter, prior to planned C1D1;
   5. Hormonal or other adjunctive therapy for cancers other than the cancer under evaluation in this study that started <14 days prior to planned C1D1 are not permitted; however, antiestrogen therapy, bisphosphonates, somatostatin analogues, leuprolide, and denosumab are permitted if started ≥14 days prior to C1D1. Other hormonal treatments and/or treatment for stable cancers (other than the cancer being treated on-study) may also be permitted 1) if these therapies would not be expected to have any positive or negative effect on the cancer being treated and 2) if discussed with and approved by the Medical Monitor;
   6. Radiation therapy <21 days prior to planned C1D1. Exception: Limited (e.g., pain palliation) radiation therapy is allowed prior to and during study drug administration as long as there are no acute toxicities, any AE due to prior radiation therapy has recovered to <Grade 2, and the radiation is not administered to a target lesion;
   7. Any prior organ transplantation, including allogeneic or autologous stem cell transplantation;
4. History of intolerance, hypersensitivity, or treatment discontinuation due to Grade 3 or greater irAEs (related to prior immunotherapy);
5. Diagnosis of immunodeficiency, either primary or acquired, or treatment with immunosuppressive levels of systemic corticosteroids (equivalent to ≥10 mg prednisone per day) or any other form of immunosuppressive therapy within 7 days prior to planned C1D1. Exception: Inhaled, intra-articular, topical, or systemic corticosteroids (systemic only at doses intended for adrenal replacement) and doses of immunosuppressive agents used prophylactically for contrast allergies are permitted in the absence of active autoimmune disease;
6. Known severe intolerance or life-threatening hypersensitivity reactions to humanized mAbs or IV immunoglobulin preparations; any history of anaphylaxis; known allergy to any of the study medications, their analogues, or excipients (sodium acetate, sucrose, sodium chloride and polysorbate 80) in the various formulations of any agent;
7. Symptomatic or uncontrolled brain metastases, leptomeningeal disease, or spinal cord compression not definitively treated with surgery or radiation (brain metastases that are stable and asymptomatic after prior treatment will be allowed);
8. Active and clinically relevant bacterial, fungal, or viral infection, including known hepatitis A, B, or C, or HIV (testing not required);
9. Women who are pregnant or breastfeeding or who plan to become pregnant/breastfeed while on study; men who plan to father children during the study;
10. History of pneumonitis requiring treatment with corticosteroids, interstitial lung disease, or severe (≥Grade 3) radiation pneumonitis (excluding localized radiation pneumonitis);
11. History in the last 3 months of acute diverticulitis, intra-abdominal abscess, or gastrointestinal obstruction, unless approved by Medical Monitor;
12. Symptomatic cardiac or cerebrovascular disease that is unresponsive to surgical or medical management;
13. Medical or social condition that, in the opinion of the Investigator, might place the subject at increased risk, adversely affect compliance, or confound safety or other clinical study data interpretation;
14. Active disease requiring systemic immunosuppressive therapy;
15. Live vaccines ≤30 days of C1D1;
16. Deep vein thrombosis, pulmonary embolism (including asymptomatic pulmonary embolism identified on imaging), or other thromboembolic event within the 6 months preceding C1D1 for JTX-8064 monotherapy cohorts only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of DLTs, treatment-emergent adverse events (TEAEs), serious TEAEs, and discontinuation due to adverse events (AEs) evaluated using National Cancer Institute (NCI) Common Technology Criteria for Adverse Events (CTCAE) version 5.0 | up to 24 months
Determination of a RP2D for JTX-8064 monotherapy and in combination with a PD-1i | up to 24 months

SECONDARY OUTCOMES:
Cmax (the maximum observed concentration) for JTX-8064 monotherapy and in combination with a PD-1i | Cycles 1 through 12 (each cycle is 21 days)
Tmax (time of maximum observed concentration) for JTX-8064 monotherapy and in combination with a PD-1i | Cycles 1 through 12 (each cycle is 21 days)
Cmin for JTX-8064 monotherapy and in combination with a PD-1i | Cycles 1 through 12 (each cycle is 21 days)
AUClast (area under the concentration-time curve from time 0 to the last measurable concentration) for JTX-8064 monotherapy and in combination with a PD-1i | Cycles 1 and 3 (each cycle is 21 days)
Cmax for PD-1i in combination with JTX-8064 | Cycles 1 through 12 (each cycle is 21 days)
Tmax for PD-1i in combination with JTX-8064 | Cycles 1 through 12 (each cycle is 21 days)
Cmin for PD-1i in combination with JTX-8064 | Cycles 1 through 12 (each cycle is 21 days)
Incidence of anti-drug antibodies (ADAs) to JTX-8064 and, as appropriate, to PD-1i | Baseline through Cycle 12 (each cycle is 21 days)
Incidence of neutralizing antibodies (Nabs) to JTX-8064 and, as appropriate, to PD-1i | Baseline through Cycle 12 (each cycle is 21 days)
For Stages 1 and 2: Receptor occupancy for LILRB2 on monocytes in whole blood | Baseline through Cycle 6 (each cycle is 21 days)
For Stages 3 and 4: Preliminary efficacy endpoints: Objective response rate (ORR; the proportion of subjects who have had a partial response [PR] or complete response [CR]) as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | up to 36 months
For Stages 3 and 4: Preliminary efficacy endpoints: Disease control rate (DCR; the proportion of subjects who have a PR, CR, or stable disease [SD]), as per RECIST version 1.1 | up to 36 months
For Stages 3 and 4: Preliminary efficacy endpoints: Progression-free survival (PFS; the interval from start of treatment to the earlier of first documentation of disease progression or death from any cause) | up to 36 months
For Stages 3 and 4: Preliminary efficacy endpoints: Overall survival (OS; the interval from start of treatment to death of any cause) | up to 36 months
For Stages 3 and 4: Preliminary efficacy endpoints: Duration of response (DOR; the time from documentation of tumor progression or death due to any cause, whichever comes first) | up to 36 months
For Stages 3 and 4: Preliminary efficacy endpoints: Percentage of subjects with tumor reduction at any time | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Stew Kroll, Study Director — Jounce Therapeutics, Inc.
Locations (45):
- United States (45):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - University of Arkansas Medical Sciences, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - California Cancer Associates for Research & Excellence, Inc., La Jolla, California
  - University of California, San Diego, La Jolla, California
  - Cedars Sinai, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - University of California, Davis, Sacramento, California
  - Yale University, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Adventist Health System/Sunbelt, Inc., Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Augusta Oncology Associates - Wheeler Road, Augusta, Georgia
  - University of Chicago, Chicago, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - University of Kentucky Chandler Medical Center (UKCMC), Lexington, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - START Midwest -Cancer & Hematology Center of Western Michigan, Grand Rapids, Michigan
  - Regents of the University of Minnesota, Minneapolis, Minnesota
  - Weill Cornell, New York, New York
  - Mount Sinai, New York, New York
  - Montefiore Medical Center PRIME, New York, New York
  - Carolina BioOncology, Huntersville, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - UC Health, LLC, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Portland Cancer Center, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Mary Crowley Cancer Research, Dallas, Texas
  - Oncology Consultants, P.A., Houston, Texas
  - MD Anderson, Houston, Texas
  - Joe Arrington Cancer Research & Treatment Center, Lubbock, Texas
  - START Texas Accelerated Research Therapeutics, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
  - The Board of Regents of the University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin